CLINICAL TRIAL: NCT00833664
Title: The Relative Bioavailability of Two Terbinafine HCl 250 mg Tablet Formulations Under Non-Fasting Conditions
Brief Title: Terbinafine HCl 250 mg Tablet Formulations Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10136025
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Terbinafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terbinafine (Experimental): Terbinafine 250 mg Tablet (test) dosed in first period followed by Lamisil® 250 mg Tablet (reference) dosed in second period
  Interventions: Drug: Terbinafine HCl 250mg tablets
- Lamisil® (Active Comparator): Lamisil® 250 mg Tablet (reference) dosed in first period followed by Terbinafine 250 mg Tablet (test) dosed in second period
  Interventions: Drug: Lamisil® 250 mg Tablets

INTERVENTIONS:
Drug: Terbinafine HCl 250mg tablets — 1 x 250 mg
  Arms: Terbinafine
Drug: Lamisil® 250 mg Tablets — 1 x 250 mg
  Arms: Lamisil®

SUMMARY:
The Purpose of this study os to evaluate the relative bioavailability of the test formulation of terbinafine tablets with an already marketed reference formulation Lamisil® (Novartis Pharmaceuticals), under post-prandial conditions in healthy, non-tobacco using male and female adult subjects.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older inclusive with a body mass index (BMI) of 30 or less.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed and dated informed consent form, which meets all criteria of current FDA regulations
* If female and of child bearing potential subjects must be prepared to abstain from sexual intercourse or use a reliable barrier method of contraception (e.g. condom, IUD) during the duration of the study. Female subjects who have used oral contraceptives within 14 days or injected hormonal contraceptives within 180 days of dosing will not be allowed to participate.

Exclusion Criteria:

* If female, pregnant, lactating or likely to become pregnant during the study.
* History of allergy or sensitivity to terbinafine, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic evidence of chronic infectious disease, system disorder ot organ dysfunction.
* Presence of gastrointestinal disease ot history of malabsorption within the last year.
* History of psychiatric disorders occuring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes. within 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addition requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
* Positive test results for drug of abuse at screening.
* Tobacco user within 90 days of the first study dose.
* Unable, or unwilling to tolerate multiple venipunctures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-01; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Ann Kennedy, M.D., Principal Investigator — Novum
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Terbinafine (Test) First: Terbinafine 250 mg Tablet (test) dosed in first period followed by Lamisil® 250 mg Tablet (reference) dosed in second period
- Lamisil® (Reference) First: Lamisil® 250 mg Tablet (reference) dosed in first period followed by Terbinafine 250 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Terbinafine (Test) First | Lamisil® (Reference) First
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout: 14 Days
Arm/Group | Terbinafine (Test) First | Lamisil® (Reference) First
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0
Period: Second Intervention
Arm/Group | Terbinafine (Test) First | Lamisil® (Reference) First
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terbinafine (Test) First | Lamisil® (Reference) First | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 6 | 10
  Black | 6 | 5 | 11
  Biracial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Terbinafine in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over144 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Terbinafine: Terbinafine 250 mg Tablet (test) dosed in either period
- Lamisil®: Lamisil® 250 mg Tablet (reference) dosed in either period
Arm/Group | Terbinafine | Lamisil®
Number analyzed (Participants) | 21 | 21
ng/mL | 906 (196) | 971 (417)
Statistical Analysis 1: Comparison: Terbinafine vs Lamisil®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 98.2, 90% CI [88.1 to 109.5] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - Terbinafine in Plasma
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 144 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Terbinafine | Lamisil®
Number analyzed (Participants) | 21 | 21
ng*h/mL | 4870 (1618) | 5953 (4170)
Statistical Analysis 1: Comparison: Terbinafine vs Lamisil®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 107.6, 90% CI [104.7 to 110.6] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant) - Terbinafine in Plasma
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 144 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Terbinafine | Lamisil®
Number analyzed (Participants) | 21 | 21
ng*h/mL | 4652 (1925) | 4835 (2795)
Statistical Analysis 1: Comparison: Terbinafine vs Lamisil®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 98.2, 90% CI [92.7 to 104.0] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.